CLINICAL TRIAL: NCT02585505
Title: Tissue Distribution of F18-FDG Labeled Autologous Bone Marrow Derived Stem Cells in Patients With Type2 Diabetes Mellitus
Brief Title: Tissue Distribution of F18-FDG Labeled ABMSCT in Patients With Type2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Anil Bhansali, Head, Dept of Endocrinology, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGI NUC MED
Record Dates: First submitted 2015-10-19; First posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous (Active Comparator): stem cells will be injected through intravenously in the subjects
  Interventions: Procedure: stem cells
- superior pancreaticoduodenal (Active Comparator): stem cells
  Interventions: Procedure: stem cells
- splenic artery (Active Comparator): stem cells will be injected through splenic in the subjects
  Interventions: Procedure: stem cells

INTERVENTIONS:
Procedure: stem cells — stem cell will be injected

SUMMARY:
Stem cells have promising potential in treating diabetes. However the therapeutic outcome in diabetic patients will profoundly depend on their delivery to pancreas. Our objective is to label stem cells with PET tracer F18-FDG to carry out in vivo cell tracking. The labeled stem cells will be given through different routes (intravenous and intraarterial)and tissue distribution studied. Patients will be followed up for the next 6 months. Glucagon stimulated C peptide will be measured at baseline and at 6 months and HOMA IR and HOMA beta will be calculated.

DETAILED DESCRIPTION:
Our objective is to label stem cells with PET tracer F18-FDG to carry out in vivo cell tracking. The labeled stem cells will be given through different routes (intravenous and intraarterial)and tissue distribution studied. Patients will be followed up for the next 6 months. Glucagon stimulated C peptide will be measured at baseline and at 6 months and HOMA IR and HOMA beta will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with type 2 diabetes mellitus between 30 and 65 years of age.

  * Duration of diabetes ≥ 5 years.
  * Failure to triple OHA in optimal doses {glimepiride (4 gm), metformin(2-2.5 gm) and pioglitazone(15mg)}.
  * Requiring insulin therapy for last six month
  * On stable doses of insulin (≥0.4 IU/kg/day, Vildagliptin, metformin (2 gm), pioglitazone (15mg) for last three months.
  * GAD antibody negative status.

Exclusion Criteria:

* Patients with type 1 diabetes mellitus or secondary diabetes
* Patients with serum creatinine > 1.5 mg/dL
* Abnormal liver function tests (defined as value of transaminases > 3 times the upper value of normal or serum bilirubin higher than normal for the reference value for the laboratory).
* History of cholecystitis/ cholelithiasis/ cholecystectomy.
* Seropositivity for HIV, HBsAg and HCV.
* History of myocardial infarction or unstable angina or any cardiovascular events in the previous 3 months.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Increase in glucagon stimulated C peptide level | 6 months